CLINICAL TRIAL: NCT01189409
Title: A Randomized, Double Blind, Double-dummy, 2-treatment, 2-period Crossover Comparison of Sennosides and Polyethylene Glycol in Treatment of Opioid-induced Constipation in Outpatients With Cancer
Brief Title: Polyethylene Glycol (PEG) Versus Sennosides Study in Opioid-Induced Constipation in Cancer Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was terminated based on results of interim analysis.
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Pippa Hawley, Principal Investigator, British Columbia Cancer Agency
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H0901329
Record Dates: First submitted 2010-03-17; First posted 2010-08-26 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Constipation; Cancer
Keywords: Constipation; Opioids; Cancer; Polyethylene glycol; Sennosides; Opioid Therapy
MeSH Terms: conditions — Constipation; Neoplasms | interventions — Phenolphthalein; Sennosides

STUDY DESIGN:
Intervention Model Description: The primary outcome will be treated as a binomial outcome, expressed as the number of successful trials out of a pre-defined number of trials n = 18. Given this, the primary outcome will be analysed via a generalized mixed effects model. The model will include: (i) fixed effects for treatment, treatment period and their interaction, (ii) fixed effects for the baseline characteristics and (iii) a random patient effect. Including the latter effect in the model will help capture the within-patient correlation among the values of the primary outcome collected in Period I and Period II for the same patient.
  All statistical analyses will be conducted using the open-source statistical software package R.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind using a dummy alternate treatment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG then Senna (Experimental): PEG in stepped bowel protocol
  Interventions: Drug: PEG then Senna
- Senna then PEG (Experimental): Stepped bowel protocol with Senna then PEG
  Interventions: Drug: Senna then PEG

INTERVENTIONS:
Drug: PEG then Senna — Stepped bowel protocol with PEG for 3 weeks followed by senna for 3 weeks. Both active treatments accompanied by placebo of alternate (lactose powder).
  Other Names: Lax-a-Day
  Arms: PEG then Senna
Drug: Senna then PEG — Stepped bowel protocol with senna for 3 weeks followed by PEG for 3 weeks. Both active treatments accompanied by placebo of alternate (lactose powder).
  Other Names: senokot
  Arms: Senna then PEG

SUMMARY:
This is a study to compare the efficacy and tolerability of two laxatives for treatment of opioid-induced constipation in adult outpatients with cancer treated at the British Columbia Cancer Pain and Symptom Management/Palliative Care clinics. Each participating patient will be randomly assigned to one of two treatment groups.

DETAILED DESCRIPTION:
One group will be started on a bowel protocol of escalating doses of sennosides, plus a dummy polyethylene glycol (lactose), and the other will receive dummy sennosides capsules (lactose) plus polyethylene glycol, with the same dosing protocol. After three weeks of one active treatment the patients will switch to the alternate active product and dummy preparation. The total duration for the study will be 6 weeks for each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient (18 years and above) with diagnosis of cancer.
2. Patient requires treatment or prevention of constipation.
3. Patient is able to communicate effectively with staff.
4. Expected prognosis more than 12 weeks.
5. On or starting opioid therapy

Exclusion Criteria:

1. Patient unable to take oral medication.
2. Allergy or previous intolerance to PEG or sennosides.
3. Lactose intolerant.
4. Contraindication to PEG or sennosides.
5. Known or suspected bowel obstruction or ileus.
6. Colostomy or ileostomy.
7. Inflammatory bowel disease.
8. Hospitalisation expected within the study period.
9. Patient unable to complete the study diary in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-06; Primary Completion 2017-12 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Hawley, FRCPC, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First 3 Weeks
Arm/Group | PEG Then Senna | Senna Then PEG
Started | 37 | 33
Completed | 19 | 23
Not Completed | 18 | 10
Period: Second 3 Weeks (Switch to 2nd Treatment)
Arm/Group | PEG Then Senna | Senna Then PEG
Started | 19 | 23
Completed | 13 | 15
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG Then Senna | Senna Then PEG | Total
Number analyzed (Participants) | 37 | 33 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 22 | 42
  >=65 years | 17 | 11 | 28
Age, Continuous [Mean (Full Range); unit: years] | 72.8 [26 to 89] | 59.2 [38 to 74] | 66 [26 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 15 | 38
  Male | 14 | 18 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Diagnosis [Count of Participants; unit: Participants]
  Lung | 4 | 6 | 10
  Breast | 9 | 4 | 13
  GI | 3 | 3 | 6
  Brain | 1 | 0 | 1
  Kidney | 1 | 0 | 1
  Prostate | 3 | 3 | 6
  Bladder | 1 | 0 | 1
  Haematological | 3 | 5 | 8
  Other | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Bowel Performance Scale (BPS)
Description: Mean values of Number of Days with Satisfactory Bowel Movements Per Days of Treatment across time by treatment, derived from the mixed effects Poisson regression model. If the BPS rating on a day was -1, 0 or +1, the patient's bowel movement on that day was deemed to be satisfactory.
Time Frame: Last 18 days of each 21 day study period
Measure: Mean (Full Range); unit: Ratio
Groups:
- Polyethylene Glycol (PEG): Those patients on PEG during either treatment period
- Sennosides: Those patients on sennosides during either treatment period
Arm/Group | Polyethylene Glycol (PEG) | Sennosides
Number analyzed (Participants) | 28 | 28
Ratio
  Period 1 | 0.659 [0 to 0.941] | 0.534 [0 to 1.0]
  Period 2 | 0.641 [0.333 to 1.0] | 0.636 [0.111 to 1.0]

2. Secondary Outcome: Patient Preference
Description: The patients will be asked to state which treatment period they prefer. Only assessed using patients who completed both arms of the study (n=28).
Time Frame: end of study (6 weeks)
Measure: Count of Participants; unit: Participants
Groups:
- Polyethylene Glycol (PEG): Participants who completed both arms of the study and preferred PEG over Senna
- Senna: Participants who completed both arms of the study and preferred Senna over PEG
- No Preference: Participants who completed both arms of the study and had no preference in treatment
Arm/Group | Polyethylene Glycol (PEG) | Senna | No Preference
Number analyzed (Participants) | 28 | 28 | 28
Participants | 13 | 13 | 2

3. Secondary Outcome: Time (in Days) to Attain an Ideal BPS Score of Goal
Description: Proportion of patients in the study population estimated to reach a BPS at goal in the first period as a function of the time (in days) from day 1, presuming they were followed for 21 days and contributed a BPS score on each of those days.
  Constipation was graded using the Victoria Bowel Performance Scale (BPS), a nine-point scale from -4 (constipation) to +4 (diarrhea) which has been validated for use in patients receiving palliative care.
Time Frame: 3 weeks (ascertained at the end of period 1)
Population: Patients with a minimum of 7 days of treatment in the first period were included in the modeling.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Polyethylene Glycol (PEG): Patients on the stepped bowel protocol with PEG accompanied by placebo alternate for the first 3 weeks.
- Senna: Patients on the stepped bowel protocol with Senna accompanied by placebo alternate for the first 3 weeks.
Arm/Group | Polyethylene Glycol (PEG) | Senna
Number analyzed (Participants) | 23 | 24
Days | 6 [4 to 13] | 8 [6 to NA] — Only the lower bound could be computed

4. Secondary Outcome: Incidence of Cramps
Description: The patients were asked to indicate any experience of cramps while on study treatment
Time Frame: Last 18 days of each 21 day study period
Population: Patients who reported incidence of cramps at least once.
Measure: Count of Participants; unit: Participants
Groups:
- Polyethylene Glycol (PEG): Patients on PEG during either treatment period
- Senna: Patients on Senna during either treatment period
Arm/Group | Polyethylene Glycol (PEG) | Senna
Number analyzed (Participants) | 70 | 70
Participants | 27 | 25

5. Secondary Outcome: Rectal Measures
Description: The patients were asked to indicate any experience of rectal bleeding or rectal pain while on study treatment
Time Frame: Last 18 days of each 21 day study period
Population: Patients who reported incidence of rectal pain or rectal bleeding at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Polyethylene Glycol (PEG) | Senna
Number analyzed (Participants) | 70 | 70
Participants
  Rectal Bleeding | 7 | 6
  Rectal Pain | 10 | 9

ADVERSE EVENTS:
Time Frame: 6 weeks (the end of the second treatment period)
Arm/Group | Polyethylene Glycol (PEG) | Senna
All-Cause Mortality (participants affected / at risk) | 0/70 | 1/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 6/70 | 7/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Polyethylene Glycol (PEG) (N=70) | Senna (N=70)
Diarrhea (Gastrointestinal disorders) | 4 | 2
Dysphagia (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cramps (Gastrointestinal disorders) | 0 | 1
Dizziness (General disorders) | 0 | 1
Allergic Reaction (Product Issues) | 1 | 0 — Lactose intolerance to placebo
(General disorders) | 1 | 0 — Unable to determine patient adverse event - patient withdrew from study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT01189409/Prot_SAP_000.pdf